CLINICAL TRIAL: NCT06506513
Title: Targeting Myosteatosis Though Physical Exercise to Treat Metabolic Dysfunction-associated Steatotic Liver Disease
Brief Title: Targeting the Skeletal Muscle to Treat Metabolic Dysfunction-associated Steatotic Liver Disease
Acronym: MYO-MASLD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Concerted Research Action (Unknown); Fonds National de la Recherche Scientifique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST-IR-01 MYO-MASLD
Record Dates: First submitted 2024-06-27; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Metabolic Dysfunction-associated Steatotic Liver Disease
Keywords: metabolic dysfunction-associated steatotic liver disease; MASLD; physical activity; myosteatosis; magnetic resonance imaging; magnetic resonance specroscopy; muscle biopsy
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Patients presenting both MASLD and an excessive muscle lipid content (myosteatosis) assessed by magnetic resonance imaging will be recruited. All patients will then be randomized in three groups corresponding to three physical activity programs of increasing intensity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): in this control group, patients will perform non-cardiovascular non-intensity training (stretching, meditation).
  Interventions: Other: Low intensity exercise training
- moderate-intensity low interval training group (Active Comparator): In this group, patients will perform moderate-intensity low interval training.
  Interventions: Other: Moderate intensity exercise training
- high-intensity interval training (Active Comparator): In this group, patients willp erform high-intensity interval training.
  Interventions: Other: High-intensity interval training

INTERVENTIONS:
Other: High-intensity interval training — High-intensity interval training
  Arms: high-intensity interval training
Other: Moderate intensity exercise training — Moderate intensity exercise training
  Arms: moderate-intensity low interval training group
Other: Low intensity exercise training — Low intensity exercise training
  Arms: control group

SUMMARY:
Muscle changes including myosteatosis are reported as highly prevalent in metabolic dysfunction-associated steatotic liver disease (MASLD). Recent studies highlighted a link between muscle fat content and liver disease severity. Conversely, MASLD histological remission though diet or metabolic surgeries is also linked to a decrease in muscle fat content. Therefore, skeletal muscle appears as a potential target to treat MASLD.

DETAILED DESCRIPTION:
In this monocenter interventional study, we will assess the impact of physical activity on muscle fat content and liver disease severity in MASLD as well as the mechanisms mediating the potential beneficial effects of exercise.

ELIGIBILITY:
Inclusion Criteria:

* confirmed MASLD at abdominal imaging
* confirmed excessive muscle lipid content at imaging
* stable weight

Exclusion Criteria:

* severe comorbidities including active malignancies, neuromuscular degenerative diseases
* contraindications to physical activity
* excessive alcohol consumption

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
the impact of physical activity on muscle and liver phenotypes | every four weeks from baseline till study completion
  the investigators will assess at baseline and every four weeks till study completion the impact of intervention on liver phenotype assessed by transient elastography and muscle phenotype assessed by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Lanthier, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (2):
- Belgium (2):
  - Cliniques universitaires Saint-Luc, Brussels
  - Centre d'investigation clinique en nutrition, Louvain-la-Neuve

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Henin G, Loumaye A, Leclercq IA, Lanthier N. Myosteatosis: Diagnosis, pathophysiology and consequences in metabolic dysfunction-associated steatotic liver disease. JHEP Rep. 2023 Nov 14;6(2):100963. doi: 10.1016/j.jhepr.2023.100963. eCollection 2024 Feb. PMID 38322420
- [Result] Henin G, Loumaye A, Deldicque L, Leclercq IA, Lanthier N. Unlocking liver health: Can tackling myosteatosis spark remission in metabolic dysfunction-associated steatotic liver disease? Liver Int. 2024 Aug;44(8):1781-1796. doi: 10.1111/liv.15938. Epub 2024 Apr 16. PMID 38623714